CLINICAL TRIAL: NCT00736788
Title: A Phase 1, Single-Centre, Randomised, Double-Blind (Within Panels), Placebo-Controlled Study to Investigate Safety, Tolerability and Pharmacokinetics of AZD1704 After Administration of Oral Single Ascending Doses in Healthy Japanese Male and Non-Fertile Female Volunteers
Brief Title: Assess Safety, Tolerability and Pharmacokinetic (PK) of AZD1704 in Healthy Japanese Male and Non-Fertile Female Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: AZD1704 has essentially similar PK profile in Japanese subjects as in Caucasians. One of the main purposes of the study has thereby been achieved.
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD, Medical Science Director, Emerging Analgesia, AstraZeneca R&D Södertälje Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0980C00005; 2008-002153-20
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteers
Keywords: AZD1704,; Japanese; Healthy; Volunteers,; Phase I study,; Single Ascending Dose; Safety,; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Four different oral dose levels of a suspension containing AZD1704
  Interventions: Drug: AZD1704
- 2 (Placebo Comparator): oral suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1704 — single dose oral suspension, 4 different dose levels
  Arms: 1
Drug: Placebo — single dose oral suspension
  Arms: 2

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of AZD1704 following single ascending doses in healthy Japanese male and non-fertile female volunteers by assessment of adverse events (AEs), vital signs (supine and standing blood pressure, pulse rate, respiratory rate and body temperature), safety laboratory variables and 12 lead electrocardiography (ECG). The secondary objectives of the study are: to investigate the subjective CNS effects of orally administered AZD1704 in healthy Japanese male and non-fertile female volunteers on a psychometric rating scale by assessment of specific adjectives (stimulated, anxious, sedated, down and high) rated on visual analogue mood scale (VAMS) and to investigate the pharmacokinetic profile of AZD1704 following single ascending doses in healthy Japanese male and non-fertile female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese males and non-fertile females, defined as first generation Japanese (both parents and grandparents are of Japanese origin, the subject is born in Japan and has not been living outside of Japan for more than 5 years) aged 20-45 years .
* Clinical normal physical findings
* BMI 19 - 27, weight 50 - 95 kg

Exclusion Criteria:

* History of somatic disease/condition or ongoing psychiatric disease/condition that may interfere with the objectives of the study.
* History of psychotic disorder among first-degree relatives.
* History of use of antipsychotic, antidepressant or anxiolytic drugs, prescribed as well as non-prescribed use.
* Smoking more than 7 cigarettes per week or consumption of more than 3 portion of snuff or equivalent per day within 30 days before administration of study drug.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability - adverse events (AEs), vital signs (supine and standing blood pressure, pulse rate, respiratory rate and body temperature), safety laboratory variables and 12 lead electrocardiography (ECG) | From dosing to follow up

SECONDARY OUTCOMES:
Pharmacodynamic VAMS scores of different adjectives (stimulated, anxious, sedated, down and high). | During residential period
Pharmacokinetic profile of AZD1704 following single ascending doses in healthy Japanese male and non-fertile female volunteers | During residential period

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, Study Director — AstraZeneca R&D Södertälje; Ulrike Lorch, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Research Site, London, United Kingdom